CLINICAL TRIAL: NCT04983992
Title: Prospective Clinical Study of Excessive Lateral Pressure Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Weihai Wendeng District Central Hospital (Unknown); Inner Mongolia Autonomous Region Hospital (Unknown); Beijing Delconi Orthopaedic Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: M2020527
Record Dates: First submitted 2021-06-27; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Excessive Lateral Pressure Syndrome
Keywords: excessive lateral pressure syndrome; patellofemoral joint; tibiofemoral joint

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lateral retinaculum of the knee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group: People suffered from excessive lateral pressure syndrome with extracapsular release of lateral retinaculum.
  Interventions: Procedure: extracapsular release of lateral retinaculum
- control group: People suffered from excessive lateral pressure syndrome with conservative treatment

INTERVENTIONS:
Procedure: extracapsular release of lateral retinaculum — A new kind of surgery releases the lateral retinaculum from outside the knee capsular, maintaining the structure of the knee capsular.
  Groups: observation group

SUMMARY:
The study of July 2021 to July 2022 to undergraduate course to see a doctor and accept the lateral retinaculum capsule of external release the prospectie study of 100 patients with follow-up, compared with preoperative and postoperative imaging data, clinical manifestations, signs, etc., to evaluate the surgical effect, at the same time of resection specimens for pathology and genetics research,To investigate the pathogenesis of lateral patella compression syndrome.

DETAILED DESCRIPTION:
Excessive Lateral Pressure Syndrome (ELPS) is a series of clinical symptoms caused by various factors, such as patella tilt, adaptive contraction of the Lateral retinaculum and unbalanced Pressure on the medial and Lateral joint surfaces of the patellofemoral. The concept was first proposed by Ficat in 1977. Patellofemoral pain syndrome has long been lumped together as widespread pregenitual pain and Patella malalignment syndrome as Patellofemoral pain due to poor Patella alignment.Kramer et al. found that the main cause of patellofemoral pain and increased pressure on the lateral patellofemoral surface was excessive pressure on the lateral retinol. Later, this view was accepted by more scholars, and lateral patellofemoral compression syndrome was gradually regarded as an independent syndrome and more studies were conducted.

In patients with lateral patella compression syndrome, early manifestations are usually pain in the soft tissues around the patella. Fulkerson et al. in 1985 found pathological changes in the nerve fibers in the lateral retinaculum through a pathological study, which is the basis for early lesions showing only pain in the soft tissues around the patella.As the disease progresses, uneven pressure on the medial and lateral facets of the patellofemoral joint will gradually lead to damage of the medial and lateral facets of the articular cartilage, eventually leading to irreversible damage of the articular cartilage and osteoarthritis.

The surgical treatment of lateral compression syndrome is varied, and in recent years, the most commonly used surgical methods include: incision lysis, percutaneous lysis, arthroscope-assisted percutaneous lysis, arthroscopic release, etc.These traditional surgical methods all have obvious complications, such as intraarticular dislocation of patella, recurrence of lateral compression due to postoperative adhesion of the support band, patellofemoral joint instability, intraarticular hematoma, etc.Although there are many surgical treatment methods for lateral compression syndrome, there is still no recognized standard treatment. Due to the fact that its effect and evaluation criteria cannot be unified, accurate horizontal comparison cannot be made among different regions and different populations.

Made by the researchers of the lateral retinaculum extracapsular release, at the same time in the release of the lateral retinaculum complete retaining articular capsule and lateral patellofemoral ligament, this procedure can obviously improve patellofemoral joint trajectory anomalies and significantly reduce joint surface pressure, at the same time reduce the surgical trauma, try to keep the original structure, can greatly reduce the postoperative complications of patellofemoral joint.

Studied in this paper in March 2021 to March 2022 to undergraduate course to see a doctor and accept the lateral retinaculum capsule of external release the prospective study of 100 patients with follow-up, compared with preoperative and postoperative imaging data, clinical manifestations, signs, etc., to evaluate the surgical effect, at the same time of resection specimens for pathology and genetics research,To investigate the pathogenesis of lateral patella compression syndrome.

Through this study, to explore the etiology, development and outcome of the disease, is helpful for the early diagnosis and treatment of the disease, avoid the irreversible injury of the patient's knee joint, greatly improve the quality of life of patients, reduce the incidence of knee replacement, and save medical resources.At the same time, the external capsule release of the lateral retinacular joint created by the present study will have a profound impact on the surgical treatment of the lateral retinacular joint.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Age <40.
  2. Normal strength line of lower limbs: no valgus or varus feet (HKA <±5°)

Exclusion Criteria:

1. Combined patella dislocation and medial retinacular injury.
2. Have a history of knee surgery, knee injury and fracture.
3. Complicated cruciate ligament injury and medial and lateral collateral ligament injury.
4. Combined knee osteoarthritis.
5. Complicated with rheumatism, rheumatoid arthritis and other types of arthritis
6. Patellar bisection, trochlear dysplasia
7. Gouty arthritis and hyperuricemia of the knee
8. Complicated meniscus injury of degree III or above
9. Incorporating lateral discoid meniscus

Ages: 10 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: Young and middle-aged sports active people
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of lesions | 2years
  The improvement of cartilage injury of patellofemoral joint and tibiofemoral joint. Two senior surgeons read the MRI separately, recording the status of lesion area. The lesion area was compared before and after surgery. Using Outerbridge Classification to evaluate the severity of cartilage injury.

SECONDARY OUTCOMES:
Pain severity change | 2years
  Using Visual Analog Pain Scale for pain evaluating pain severity.The score ranks from 0 to 10. 0 means "no pain", 10 means "the pain is intolerable". The higher the score, the more pain the patient suffers.
Clinical symptom change | 2years
  Using Kujala score for symptom change.

IPD SHARING:
Plan to Share IPD: No